CLINICAL TRIAL: NCT02218242
Title: A Single-arm, Phase II Study of Thoracoscopic Lung Cancer Staging With the Use of Intraoperative Ultrasound at the Time of Definitive Resection
Brief Title: Thoracoscopic Lung Cancer Staging With the Use of Intraoperative Ultrasound
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll enough participants
Sponsor: Joel Thompson, PhD (Other)
Responsible Party: Sponsor-Investigator, Joel Thompson, PhD, Compliance Administrator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-LUN-95-MCC
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
Keywords: Lung; Cancer; Ultrasound; Staging
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ultrasound (Experimental): Participants in this study have elected to have surgical resection of non-small cell lung cancer tumors as part of their standard of care. During that surgical procedure, participants will also receive laparoscopic intraoperative ultrasound to assess the thoracic wall lymph nodes as part of the experimental procedure. The ultrasound procedure will add about 15 minutes to the total surgical time. Because it is laparoscopic and utilizes non-ionizing radiation, the risk to the participant is minimal.
  Interventions: Device: Intraoperative ultrasound

INTERVENTIONS:
Device: Intraoperative ultrasound — Intraoperative ultrasound will be performed at the completion of the standard lung cancer resection with mediastinal lymph node dissection. This evaluation will be performed by a different surgeon from the primary surgeon performing the operation to minimize operator variability with the ultrasound system and help control for bias. Additional lymph nodes identified will be resected and sent for pathologic evaluation. It is anticipated that this additional evaluation and treatment should take no more than 30 minutes and as such a time limit of 30 minutes from introduction of the ultrasound probe into the surgical field will be set.
  Other Names: B-K Medical/Analogic 8666-Radio Frequency laparoscopic ultrasound transducer and the bedside flex Focus 1202 imaging system

SUMMARY:
All patients undergoing video-assisted thoracoscopic (VATS) resection of lung cancer will receive standard therapy including lobectomy or sub-lobar resection and mediastinal lymph node dissection. After completion of the standard of care, intraoperative ultrasound will be used to evaluate lymph node stations for the presence of any missed lymph nodes with particular focus on lymph nodes which may appear pathologic on ultrasound evaluation. Data will be reviewed for rates of pathologic upstaging, and sensitivity and specificity of ultrasound as an additional diagnostic tool in the operating room will be evaluated. It is hypothesized that Intra-operative thoracoscopic ultrasound following standard video-assisted thoracoscopic (VATS) dissection will increase the rate of pathologically staged in N2 nodes in non-small cell lung cancer patients undergoing definitive surgical resection.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years. Eastern Cooperative Oncology Group performance status ≤2 (Karnofsky ≥60%, see Appendix A).

Life expectancy of greater than 3 months

Patients be able to undergo VATS resection as defined below:

* Preoperative Forced Expiratory Volume at one second ≥ 40% predicted
* OR
* Post-operative predicted Forced Expiratory Volume at one second ≥ 0.8 l
* Hg ≥ 8.0
* No evidence of coronary ischemia on stress evaluation Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Patients with surgery for a prior ipsilateral lung cancer

Patients with known brain metastases

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. (Patients with HIV are not excluded from this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Thompson, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Markey Cancer Center, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound: Intraoperative ultrasound
  Intraoperative ultrasound: Intraoperative ultrasound
Period: Overall Study
Arm/Group | Ultrasound
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants] — Age information was collected at the time of consenting
  Participants
    <=18 years | 0
    Between 18 and 65 years | 3
    >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Detection of Occult Pathologic N2 Lymph Nodes
Description: Participants undergoing resection of lung tumors will have laparoscopic thoracic wall ultrasound in an attempt to identify pathologic N2 lymph nodes. Data will be presented as the ratio of lymph nodes identified as cancerous to the total number of lymph nodes investigated with the ultrasound technique.
Time Frame: At time of surgery
Population: An insufficient number of participants were consented to generate meaningful data for this study. We reached an enrollment of less than 10% of what our power calculations suggested we needed. No pathologic lymph nodes were identified, thus the percent of pathologic lymph nodes is in fact zero
Measure: Number; unit: percentage of pathologic lymph nodes
Units Other Than Participants: lymph nodes
Arm/Group | Ultrasound
Number analyzed (Participants) | 9
Number analyzed (lymph nodes) | 20
percentage of pathologic lymph nodes | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected in the operating room at the time of the procedure. Typically less that 30 minutes.
Description: Patients were assessed for adverse events through investigator assessment at the time of the procedure
Arm/Group | Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
The University of Kentucky Medical Center did not treat a sufficient patient population to enroll and complete this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT02218242/Prot_SAP_000.pdf